CLINICAL TRIAL: NCT00691795
Title: Comparison of Fentanyl-bupivacaine and Clonidine-bupivacaine for Breakthrough Pain in Advanced Labor in Patients With Continuous Epidural Analgesia
Brief Title: Epidural Fentanyl-bupivacaine Versus Clonidine-bupivacaine for Breakthrough Pain in Advanced Labor
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was recently terminated due to poor enrollment - never enrolled.
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAC9826
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Labor Pain
Keywords: Analgesia; Epidural; Pregnancy; Labor; Clonidine; Fentanyl; Bupivacaine; Childbirth
MeSH Terms: conditions — Labor Pain; Agnosia | interventions — Clonidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CLONIDINE (Experimental): Participants randomized to this arm of the study receive 75 micrograms clonidine with the bupivacaine in their epidural when requesting pain relief in advanced labor
  Interventions: Drug: Clonidine or fentanyl
- FENTANYL (Experimental): Participants randomized to this arm of the study receive 75 micrograms fentanyl with the bupivacaine in their epidural when requesting pain relief in advanced labor
  Interventions: Drug: Clonidine or fentanyl

INTERVENTIONS:
Drug: Clonidine or fentanyl — After obtaining consent, the patients will be randomized into two groups using a random allocation table. At the onset of late stage breakthrough pain one arm of patients will receive a mixture of 75 mcg clonidine and 10 mg bupivacaine in 8 ml of volume and the second group will receive 75 mcg fentanyl and 10 mg bupivacaine in 8 ml of volume.
  Other Names: Clonidine = "DuraClon"; Fentanyl= fentanyl = Sublimaze

SUMMARY:
Epidural analgesia is widely regarding as the most effective analgesic strategy for labor pain. Modern practice is to utilize dilute local anesthetics as a continuous infusion along with an opioid, e.g., our common "recipe" of 12 ml/hr of 0.0625% bupivacaine with 2 micrograms/ml fentanyl, after the initial dose to maintain patient comfort until delivery. This dose of the infusion often provides adequate comfort without interfering with the mobility of the patient and her ability to effectively push during delivery. However, this low dose epidural infusion strategy often results in recurrence of pain after an initial pain free period.

This breakthrough pain is treated by administering small boluses of analgesics via the epidural catheter. The pain occurring in labor is initially of visceral origin and is mediated by pain fibers originating from the low thoracic and upper lumbar segments of the spinal cord. As labor progresses to the late first phase (also known as transitional stage), pain sensations originating from the distension of the pelvic floor, vagina and perineum adds a somatic component to labor pain. This type of breakthrough pain is often difficult to treat.

Although requests from patients to alleviate late stage breakthrough pain are common, no one knows the most effective strategy for pain management in this stage of labor. This study is designed to compare the efficacy of two treatments for controlling late first stage breakthrough pain during labor with an epidural infusion in place: clonidine-bupivacaine versus fentanyl-bupivacaine.

Women who have labor epidural analgesia in place will be enrolled to be randomized if and when they present with breakthrough pain in the late first stage or second stage of labor (≥ 8 cm dilated). They will receive 8 ml of a solution containing 10 mg bupivacaine and 75 micrograms of either fentanyl (an opioid or "narcotic") or clonidine (an "alpha-2 agonist known to be effective as an epidural analgesic).

Pain relief, labor progress and outcome will be assessed to compare fentanyl versus clonidine.

It is the hypothesis of this study that clonidine added to bupivacaine is a better analgesic than fentanyl added to bupivacaine for breakthrough pain in advanced labor.

ELIGIBILITY:
Inclusion Criteria:

* women in labor at term pregnancy
* healthy
* epidural analgesia in place
* breakthrough pain in advanced labor

Exclusion Criteria:

* chronic pain syndrome
* receiving systemic opioids within 4 hours
* receiving chronic antidepressants, clonidine, opioids

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pain score on a VAS scale (success = score less than or equal to 2 on a 10 point scale) | 15 minutes

SECONDARY OUTCOMES:
Maternal blood pressure | 2 hours
Maternal heart rate | 2 hour
Neonatal Apgar score | 1 and 5 minutes post delivery
Mode of delivery (spontaneous vaginal versus instrumental vaginal versus cesarean | at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Smiley, MD, Principal Investigator — Professor of Clinical Anesthesiology, Columbia University; Imre Redai, MD, Principal Investigator — Assistant Professor, Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States